CLINICAL TRIAL: NCT01261312
Title: A Phase 1-2, Dose Escalation, Multicenter Study of Two Subcutaneous Regimens of SGI-110, a DNA Hypomethylating Agent, in Subjects With Intermediate or High-Risk Myelodysplastic Syndromes (MDS) or Acute Myelogenous Leukemia (AML)
Brief Title: SGI-110 in Participants With Myelodysplastic Syndromes (MDS) or Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SGI-110-01
Record Dates: First submitted 2010-11-29; First posted 2010-12-16 (Estimated); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: MDS; CMML; AML
Keywords: SGI-110; DNA Hypomethylating Agent; Intermediate 1, Intermediate 2, CMML or High Risk MDS; AML
MeSH Terms: interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily (Experimental): Participants received starting dose of guadecitabine 3 milligrams per meter square (mg/m^2), subcutaneously (SC), daily from Days 1-5, of a 28-day cycle. The dose was subsequently increased to 9, 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
  Interventions: Drug: Guadecitabine
- Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly (Experimental): Participants received starting dose of guadecitabine 6 mg/m^2, SC, once weekly on Days 1, 8 and 15, of a 28-day cycle. The dose was subsequently increased to 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
  Interventions: Drug: Guadecitabine
- Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly (Experimental): Participants received starting dose of guadecitabine 60 mg/m^2, SC, twice weekly on Days 1, 4, 8, 11, 15 and 18, of a 28-day cycle. The dose was subsequently increased to 90 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
  Interventions: Drug: Guadecitabine
- Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 60 mg/m^2, SC, daily, from Days 1-5, of a 28-day cycle in participants with diagnosis relapsed/refractory (r/r) AML.
  Interventions: Drug: Guadecitabine
- Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 90 mg/m^2, SC, daily, from Days 1-5, of a 28-day cycle in participants with a diagnosis of r/r AML.
  Interventions: Drug: Guadecitabine
- Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) (Experimental): Participants received guadecitabine 60 mg/m^2, SC, daily from Days 1-5 and 8-12, of a 28-day cycle in participants with a diagnosis of r/r AML.
  Interventions: Drug: Guadecitabine
- Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 60 mg/m^2, SC, daily from Days 1-5, SC of a 28-day cycle in participants with a diagnosis of treatment naïve (TN) AML.
  Interventions: Drug: Guadecitabine
- Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 90 mg/m^2, SC, daily, from Days 1-5, of a 28-day cycle in participants with a diagnosis of TN AML.
  Interventions: Drug: Guadecitabine
- Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) (Experimental): Participants received guadecitabine 60 mg/m^2, SC, daily from Days 1-5 and 8-12, of a 28-day cycle in participants with a diagnosis of TN AML.
  Interventions: Drug: Guadecitabine
- Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 60 mg/m^2, SC, daily on Days 1-5, of a 28-day cycle in participants with a diagnosis of r/r Myelodysplastic Syndromes (MDS).
  Interventions: Drug: Guadecitabine
- Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 90 mg/m^2, SC, daily on Days 1-5, of a 28-day cycle in participants with a diagnosis of r/r MDS.
  Interventions: Drug: Guadecitabine
- Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 60 mg/m^2, SC, daily on Days 1-5, of a 28-day cycle in participants with a diagnosis of TN MDS.
  Interventions: Drug: Guadecitabine
- Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day) (Experimental): Participants received guadecitabine 90 mg/m^2, SC daily on Days 1-5, of a 28-day cycle in participants with a diagnosis of TN MDS.
  Interventions: Drug: Guadecitabine

INTERVENTIONS:
Drug: Guadecitabine — Subcutaneous injection
  Other Names: SGI-110

SUMMARY:
Phase 1-2 dose-escalation randomized study in participants with intermediate or high risk myelodysplastic syndromes (MDS) or acute myelogenous leukemia (AML). The Dose Escalation Segment will evaluate the biological activity, preliminary safety and efficacy of SGI-110 with two dosing schedules in MDS and AML participants while the Dose Expansion Segment will further evaluate safety and efficacy at the biological effective dose (BED) or maximum tolerated dose (MTD) as defined in the Dose Escalation Segment.

DETAILED DESCRIPTION:
Once the biologically effective dose (BED) and maximum tolerated dose (MTD) is determined in the Dose Escalation Segment, the Dose Expansion Segment will randomize participants with MDS, treatment naïve elderly acute myeloid leukemia (AML), and relapsed/refractory AML participants to receive the BED or MTD dose. Relapsed/refractory AML participants may also receive SGI-110 on a daily x 10 schedule based on the total dose per cycle evaluated in the Dose-escalation Segment using the 5-daily regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 18 years of age or older, with a confirmed diagnosis of international prognostic scoring system (IPSS) intermediate-1, intermediate-2 or high-risk MDS including Chronic Myelomonocytic Leukemia (CMML) or AML.

   * In the Dose Escalation Segment, participants who are refractory, relapsed, or unresponsive to standard treatment.
   * In the Dose Expansion Segment, hypomethylating agent (HMA) treatment-naïve MDS participants (including CMML), and intermediate-2 or high-risk MDS participant (including CMML) relapsed or refractory to prior HMA treatment are allowed, and treatment-naïve AML participants who is at least 65 years of age will be allowed if they also have at least one of the following criteria

     * AML secondary to MDS, chemotherapy, or radiation therapy
     * poor cytogenetics
     * pre-existing clinically significant dysfunction of the heart or Chronic Obstructive Pulmonary Disease (COPD)
     * poor performance status, Eastern Cooperative Oncology Group (ECOG), of 2
2. Eastern ECOG performance status of 0 to 2.
3. Adequate organ function.
4. Prior allogeneic stem cell transplant, no evidence of active graft-versus host disease (GVHD) and must be ≥ 2 weeks off immunosuppressive therapy.
5. No major surgery within 4 weeks of first dose of SGI-110.
6. No chemotherapy within 2 weeks of first dose of SGI-110 (minimum of 6 weeks for nitrosoureas and 8 weeks for bone marrow transplantation) with the exception of hydroxyurea which will be allowed during course 1 of treatment.
7. Sign an approved informed consent form for this study.

Exclusion Criteria:

1. In the Dose Expansion Segment, which includes the 10-day regimen, participants who have received 2 complete full dose cycles or more of a hypomethylating agent (HMA) decitabine or azacitidine (except for intermediate-2 or high-risk MDS participant (including CMML) relapsed or refractory to prior HMA treatment).
2. Acute promyelocytic leukemia (M3 classification).
3. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the participant has been disease free for at least 3 years.
4. Life-threatening illnesses other than AML or MDS, uncontrolled medical conditions or organ system dysfunction which, in the investigator's opinion, could compromise the participant's safety, or put the study outcomes at risk.
5. Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).
6. Hypersensitivity to decitabine, SGI-110, or SGI-110 excipients.
7. With the exception of treatment-naïve elderly AML participants, participants with uncontrolled congestive heart failure (CHF), coronary heart disease (CAD), chronic obstructive pulmonary disease (COPD), or left ventricular ejection fraction (LVEF) of ≤ 50% are excluded, symptomatic or uncontrolled arrhythmias or on continuous corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2016-07-22 (Actual); Study Completion 2016-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (15):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - University of Chicago Cancer Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chung W, Kelly AD, Kropf P, Fung H, Jelinek J, Su XY, Roboz GJ, Kantarjian HM, Azab M, Issa JJ. Genomic and epigenomic predictors of response to guadecitabine in relapsed/refractory acute myelogenous leukemia. Clin Epigenetics. 2019 Jul 22;11(1):106. doi: 10.1186/s13148-019-0704-3. PMID 31331399
- [Derived] Garcia-Manero G, Roboz G, Walsh K, Kantarjian H, Ritchie E, Kropf P, O'Connell C, Tibes R, Lunin S, Rosenblat T, Yee K, Stock W, Griffiths E, Mace J, Podoltsev N, Berdeja J, Jabbour E, Issa JJ, Hao Y, Keer HN, Azab M, Savona MR. Guadecitabine (SGI-110) in patients with intermediate or high-risk myelodysplastic syndromes: phase 2 results from a multicentre, open-label, randomised, phase 1/2 trial. Lancet Haematol. 2019 Jun;6(6):e317-e327. doi: 10.1016/S2352-3026(19)30029-8. Epub 2019 May 3. PMID 31060979
- [Derived] Issa JJ, Roboz G, Rizzieri D, Jabbour E, Stock W, O'Connell C, Yee K, Tibes R, Griffiths EA, Walsh K, Daver N, Chung W, Naim S, Taverna P, Oganesian A, Hao Y, Lowder JN, Azab M, Kantarjian H. Safety and tolerability of guadecitabine (SGI-110) in patients with myelodysplastic syndrome and acute myeloid leukaemia: a multicentre, randomised, dose-escalation phase 1 study. Lancet Oncol. 2015 Sep;16(9):1099-1110. doi: 10.1016/S1470-2045(15)00038-8. Epub 2015 Aug 19. PMID 26296954

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 94 participants with Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndromes (MDS) were enrolled in Dose escalation Phase 1, out of which 93 received treatment; Total 108 participants with relapsed and refractory (r/r) AML were enrolled, and 103 received study treatment; 107 participants with TN AML were enrolled, and 103 participants received study treatment; 105 participants with MDS were enrolled, and 102 received study treatment in Dose expansion (DE) Phase 2.
Groups:
- Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily: Participants received starting dose of guadecitabine 3 milligrams per meter square (mg/m^2), subcutaneously (SC), daily from Days 1-5 of a 28-day cycle. The dose was subsequently increased to 9, 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
- Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly: Participants received starting dose of guadecitabine 6 mg/m^2, SC, once weekly on Days 1, 8 and 15 of a 28-day cycle. The dose was subsequently increased to 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
- Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly: Participants received starting dose of guadecitabine 60 mg/m^2, SC, twice weekly on Days 1, 4, 8, 11, 15 and 18 of a 28-day cycle. The dose was subsequently increased to 90 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
- Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily,from Days 1-5 of a 28-day cycle in participants with diagnosis of relapsed/refractory (r/r) AML.
- Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day): Participants received guadecitabine 90 mg/m^2, SC, daily, from Days 1-5of a 28-day cycle in participants with a diagnosis of r/r AML.
- Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day): Participants received guadecitabine 60 mg/m^2, SC, daily from Days 1-5 and 8-12of a 28-day cycle in participants with a diagnosis of r/r AML.
- Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, dailyfrom Days 1-5, SC of a 28-day cycle in participants with a diagnosis of treatment naïve (TN) AML.
- Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day): Participants received guadecitabine 90 mg/m^2, SC, daily, from Days 1-5of a 28-day cycle in participants with a diagnosis of TN AML.
- Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day): Participants received guadecitabine 60 mg/m^2, SC, daily, from Days 1-5 and 8-12of a 28-day cycle in participants with a diagnosis of TN AML.
- Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily on Days 1-5 of a 28-day cycle in participants with a diagnosis of r/r Myelodysplastic Syndromes (MDS).
- Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day): Participants received guadecitabine 90 mg/m^2, SC, daily on Days 1-5of a 28-day cycle in participants with a diagnosis of r/r MDS.
- Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily on Days 1-5 of a 28-day cycle in participants with a diagnosis of TN MDS.
- Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day): Participants received guadecitabine 90 mg/m^2, SC. daily on Days 1-5 of a 28-day cycle in participants with a diagnosis of TN MDS.
Period: Dose Escalation Phase (Day 0- Week 170)
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Started | 44 | 35 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Data Set (Participants who received at least one dose of study treatment were included in safety data set.) | 44 | 34 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 44 | 35 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 27 | 26 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Withdrew Consent | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Hematopoietic Cell Transplant (HCT) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: DE Phase: r/r AML (Week 75-242)
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Started | 0 | 0 | 0 | 25 | 28 | 55 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Data Set (Participants who received at least one dose of study treatment were included in safety data set.) | 0 | 0 | 0 | 24 | 26 | 50 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 24 | 27 | 55 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 14 | 16 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 4 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HCT | 0 | 0 | 0 | 5 | 3 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: DE Phase: TN AML (Week 85-283)
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 28 | 53 | 0 | 0 | 0 | 0
Safety Data Set (Participants who received at least one dose of study treatment were included in safety data set.) | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 27 | 52 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 26 | 50 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 11 | 17 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 11 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 9 | 0 | 0 | 0 | 0
Not completed — Bone marrow (BM)/Stem cell transplant | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 6 | 0 | 0 | 0 | 0
Period: DE Phase: r/r MDS &TN MDS (Week 78-298)
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 27 | 28 | 23
Safety Data Set (Participants who received at least one dose of study treatment were included in safety data set.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 27 | 27 | 22
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 25 | 27 | 20
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 9 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 3 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 2
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 3 | 5
Not completed — BM/Stem Cell Transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 6 | 4
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Efficacy data set included all participants who received at least one dose of study drug.
Groups:
- Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily: Participants received starting dose of guadecitabine 3 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle. The dose was subsequently increased to 9, 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
- Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly: Participants received starting dose of guadecitabine 6 mg/m^2, SC, once weekly on Days 1, 8 and 15of a 28-day cycle. The dose was subsequently increased to 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
- Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly: Participants received starting dose of guadecitabine 60 mg/m^2, SC, twice weekly on Days 1, 4, 8, 11, 15 and 18of a 28-day cycle. The dose was subsequently increased to 90 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
- Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily,from Days 1-5 of a 28-day cycle in participants with diagnosis of r/r AML.
- Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily from Days 1-5, SC of a 28-day cycle in participants with a diagnosis of TN AML.
- Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily on Days 1-5 of a 28-day cycle in participants with a diagnosis of r/r MDS.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day) | Total
Number analyzed (Participants) | 44 | 34 | 15 | 24 | 26 | 53 | 24 | 27 | 52 | 26 | 27 | 27 | 22 | 401
Age, Continuous [Mean (Full Range); unit: years] | 66.22 [36.7 to 86.1] | 64.90 [29.1 to 83.4] | 71.04 [51.4 to 84.6] | 55.83 [22.0 to 77.0] | 62.01 [30.0 to 81.7] | 58.86 [29.2 to 82.5] | 77.83 [62.0 to 92.5] | 78.46 [66.7 to 92.6] | 77.78 [66.4 to 92.3] | 71.61 [54.7 to 85.5] | 72.05 [51.9 to 88.7] | 68.38 [18.1 to 85.3] | 71.27 [63.8 to 84.5] | 68.94 [18.1 to 92.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 3 | 9 | 6 | 26 | 10 | 11 | 18 | 10 | 11 | 6 | 8 | 145
  Male | 25 | 26 | 12 | 15 | 20 | 27 | 14 | 16 | 34 | 16 | 16 | 21 | 14 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 5 | 3 | 5 | 2 | 0 | 1 | 0 | 2 | 3 | 1 | 29
  Not Hispanic or Latino | 42 | 32 | 12 | 19 | 23 | 48 | 22 | 27 | 51 | 26 | 25 | 24 | 21 | 372
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 2 | 4 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Black or African American | 2 | 3 | 1 | 4 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 16
  White | 39 | 31 | 14 | 18 | 21 | 44 | 23 | 24 | 50 | 25 | 25 | 25 | 22 | 361
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase- Biological Effective Dose (BED): Percent Change From Baseline in DNA Long Interspersed Nucleotide Element-1 (LINE-1) Demethylation
Description: DNA LINE-1 demethylation is defined as the largest percent decrease from baseline in methylation values within a participant between Day 8 and Day 22 of the first treatment cycle. BED was assessed based on DNA LINE-1 demethylation results and defined as the smallest dose that achieves the maximum biological pharmacodynamic (PD) effect (LINE-1 demethylation) in at least 3 successive dose levels.
Time Frame: Cycle 1 Day 8
Population: Pharmacodynamic (PD) analysis set included all participants who provided evaluable blood samples for analysis of at least one PD parameter or biomarker being tested. Overall number analyzed is number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 30 | 28 | 11
percent change | -16.143 (12.692) | -4.362 (5.484) | -10.574 (8.444)

2. Primary Outcome: Dose Escalation Phase- Biological Effective Dose (BED): Percent Change From Baseline in DNA Long Interspersed Nucleotide Element-1 (LINE-1) Demethylation
Description: as for outcome 1
Time Frame: Cycle 1 Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 26 | 29 | 12
percent change | -10.359 (9.837) | -5.312 (5.796) | -17.540 (9.207)

3. Primary Outcome: Dose Escalation Phase- Biological Effective Dose (BED): Percent Change From Baseline in DNA Long Interspersed Nucleotide Element-1 (LINE-1) Demethylation
Description: as for outcome 1
Time Frame: Cycle 1 Day 22
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 30 | 22 | 8
percent change | -6.325 (7.477) | -4.777 (4.765) | -16.959 (10.112)

4. Primary Outcome: Dose Escalation Phase- Biological Effective Dose (BED): Percent Change From Baseline in DNA Long Interspersed Nucleotide Element-1 (LINE-1) Demethylation
Description: as for outcome 1
Time Frame: Cycle 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 24 | 19 | 5
percent change | -2.805 (4.249) | -1.860 (3.844) | -13.346 (6.039)

5. Primary Outcome: Dose Escalation Phase-Maximum Tolerated Dose (MTD): Number of Participants With Dose Limiting Toxicity (DLT)
Description: The MTD was defined as the largest dose for which less than 33% of subjects experienced a dose limiting toxicity (DLT) during Cycle 1 of guadecitabine administration at each dose level. DLTs were defined using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0).
Time Frame: From the start of study treatment up to 30 days post treatment (Up to approximately 46 months)
Population: Safety data analysis set included all regimen 1, 2A and 2 B participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 44 | 34 | 15
Participants
  DLT | 2 | 0 | 0
  Adverse Event (AE) | 44 | 34 | 15

6. Primary Outcome: Dose Expansion (DE) Phase- r/r AML, TN AML: Composite Complete Response (CRc) Rate
Description: Composite complete response (CRc) rate is defined as the percentage of participants whose best response is complete remission [CR], CR with incomplete platelet recovery [CRp], or CR with incomplete hematological recovery [CRi]) after treatment with study drug. CR as per AML response criteria is defined as peripheral blood absolute neutrophil count (ANC) ≥1.0×10^9/L, Platelets ≥100×10^9/L, independence from red blood cell (RBC) and platelet transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRp as per AML response criteria is defined as peripheral blood ANC ≥1.0×10^9/L, Platelets <100×10^9/L, independence from RBC transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRi as per AML response criteria is defined as peripheral blood ANC <1.0×10^9/L, no myeloblasts and <5% myeloblasts in bone marrow.
Time Frame: At end of each Cycle of 28 days (Up to approximately 38 months)
Population: Efficacy analysis set included r/r AML and TN AML participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day): Participants received guadecitabine 60 mg/m^2, SC, daily, from Days 1-5 of a 28-day cycle in participants with diagnosis of r/r AML.
Arm/Group | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day)
Number analyzed (Participants) | 24 | 26 | 53 | 24 | 27 | 52
percentage of participants | 12.5 [2.7 to 32.4] | 19.2 [6.6 to 39.4] | 30.2 [18.3 to 44.3] | 54.2 [32.8 to 74.4] | 59.3 [38.8 to 77.6] | 50.0 [35.8 to 64.2]

7. Primary Outcome: Dose Expansion (DE) Phase- r/r MDS, TN MDS: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with complete response(CR), partial response(PR), marrow complete response(mCR) and haematological improvement(HI). CR:normal peripheral counts with persistent granulocyte count ≥1.0×10^9/L, platelet count ≥100×10^9/L and normal bone marrow (BM) with persistent marrow blasts ≤5%; persistent dysplasia was noted. PR:normal peripheral counts with granulocyte count ≥1.0×10^9/L and platelet count ≥100 ×10^9/L and normal BM with marrow blasts >5% but were reduced by 50% or more. mCR:reduction of BM blasts to ≤5% without normalization of peripheral counts. HI is divided as erythroid response(HI-E): hemoglobin increase ≥1.5 g/dL or red blood cells transfusion independence, platelet response (HI-P): absolute increase of platelet count from <20 to >20×10^9/L and by at least 100%,/if more than 20×10^9/L, by an absolute increase of 30×10^9/L, neutrophil response (HI-N): granulocyte increase ≥100%, and by an absolute increase ≥0.5×10^9/L.
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included r/r MDS and TN MDS participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 26 | 27 | 27 | 22
percentage of participants | 31 [14.3 to 51.8] | 56 [35.3 to 74.5] | 48 [28.7 to 68.1] | 55 [32.2 to 75.6]

8. Secondary Outcome: Dose Escalation Phase: Response Rate in AML Participants
Description: Response rate for AML participants was assessed by Modified International Working Group (IWG) 2003 response criteria with complete response (CR), complete response with incomplete platelet recovery (CRp), CR with incomplete blood count recovery(CRi), and partial response (PR). CR: absolute neutrophil count (ANC) >1.0×10^9/L, platelets ≥100×10^9/L, independence from RBC and platelet transfusions, no or <5% myeloblasts in bone marrow(BM). CRp: ANC >1.0×10^9/L, Platelets <100×10^9/L, independence from RBC transfusions, no or <5% myeloblasts in BM. CRi: ANC <1.0×10^9/L, no or <5% myeloblasts in BM. PR: ANC >1.0×10^9/L, Platelets ≥100×10^9/L, no or decrease of ≥50% in myeloblasts to 5-25% in BM.
Time Frame: At end of each Cycle of 28 days (Up to approximately 23 months)
Population: Efficacy analysis set included regimen 1, 2A and 2B participants who received at least one dose of study drug. Overall number of participants analyzed are the number of participants with AML available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 35 | 28 | 11
percentage of participants | 11.4 [3.2 to 26.7] | 7.1 [0.9 to 23.5] | 0.0 [0.0 to 28.5]

9. Secondary Outcome: Dose Escalation Phase: Response Rate in MDS Participants
Description: Response rate for MDS participants was assessed by IWG 2006 Response Criteria with CR, PR, marrow complete response(mCR) and HI. CR: normal peripheral counts with persistent granulocyte count ≥1.0×10^9/L, platelet count ≥100×10^9/L; normal BM with persistent marrow blasts ≤5%; persistent dysplasia. PR: Normal peripheral counts with granulocyte count ≥1.0×10^9/L, platelet count ≥100×10^9/L and normal BM with blasts >5% but reduced by 50% or more. mCR: reduction of BM blasts to ≤5% without normalization of peripheral counts.
Time Frame: At end of each Cycle of 28 days (Up to approximately 23 months)
Population: Efficacy analysis set included regimen 1, 2A and 2B participants who received at least one dose of study drug. Overall number of participants analyzed are the number of participants with MDS available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 9 | 6 | 4
percentage of participants | 22.2 [2.8 to 60.0] | 50.0 [11.8 to 88.2] | 25.0 [0.6 to 80.6]

10. Secondary Outcome: Dose Escalation and Dose Expansion Phase- r/r AML, TN AML: Duration of Response
Description: Duration of response (in number of days) was calculated from the first time a complete response (CR, CRp, or CRi) was observed to time of relapse defined as the earliest time point whereby BM blasts or peripheral blood blasts become ≥5% and stayed at that level in subsequent visits while participants were still on study. CR:normal peripheral counts with persistent granulocyte count ≥1.0×10^9/L, platelet count ≥100×10^9/L and normal bone marrow (BM) with persistent marrow blasts ≤5%; persistent dysplasia was noted. CRp as per AML response criteria is defined as peripheral blood ANC ≥1.0×10^9/L, Platelets <100×10^9/L, independence from RBC transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRi as per AML response criteria is defined as peripheral blood ANC <1.0×10^9/L, no myeloblasts and <5% myeloblasts in bone marrow.
Time Frame: At end of each Cycle of 28 days (Up to approximately 38 months)
Population: Efficacy analysis set included regimen 1, 2A and 2B, r/r AML and TN AML participants who received at least one dose of study drug. Data for responders was reported for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day)
Number analyzed (Participants) | 4 | 2 | 0 | 3 | 5 | 16 | 13 | 16 | 26
days | 213.0 [47 to 350] | 300.0 [42 to 558] |  | 816.0 [15 to 880] | 112.0 [55 to 879] | 233.0 [42 to 898] | 237.0 [8 to 1068] | 185.5 [16 to 948] | 269.5 [40 to 669]

11. Secondary Outcome: Dose Escalation Phase: Hematologic Improvement Rate in MDS
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included regimen 1, 2A and 2B participants who received at least one dose of study drug. Overall number of participants analyzed are the number of participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 9 | 6 | 4
percentage of participants | 0.0 [0.0 to 33.6] | 50.0 [11.8 to 88.2] | 25.0 [0.6 to 80.6]

12. Secondary Outcome: DE Phase- r/r MDS, TN MDS: Duration of Response
Description: DOR was calculated from first time a response category (CR, PR, mCR, or HI) was achieved until response category was no longer met or the last available time point, whichever occurred first. CR:normal peripheral counts with persistent granulocyte count ≥1.0×10^9/L, platelet count ≥100×10^9/L and normal bone marrow (BM) with persistent marrow blasts ≤5%; persistent dysplasia was noted. PR:normal peripheral counts with granulocyte count ≥1.0×10^9/L and platelet count ≥100 ×10^9/L and normal BM with marrow blasts >5% but were reduced by 50% or more. mCR:reduction of BM blasts to ≤5% without normalization of peripheral counts. HI is divided as erythroid response(HI-E): hemoglobin increase ≥1.5 g/dL or RBC transfusion independence, platelet response (HI-P): absolute increase of platelet count from <20 to >20×10^9/L by at least 100%,/if more than 20×10^9/L, by absolute increase of 30×10^9/L, neutrophil response (HI-N): granulocyte increase ≥100%, by an absolute increase ≥0.5×10^9/L.
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included participants with MDS who received at least one dose of study drug. Overall number of participants analyzed are the number of participants with response. Number analyzed are the number of participants with data available for analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 6 | 12 | 12 | 11
days
  CR+PR+mCR: number analyzed (Participants) | 5 | 12 | 7 | 11
  CR+PR+mCR | 295.0 [101 to 529] | 207.0 [42 to 984] | 103.0 [35 to 1144] | 165.0 [42 to 958]
  HI: number analyzed (Participants) | 6 | 9 | 12 | 9
  HI | 202.5 [91 to 574] | 193.0 [71 to 1050] | 227.0 [89 to 525] | 127.0 [81 to 1087]

13. Secondary Outcome: Dose Escalation r/r AML, TN AML: Time to Response
Description: Time to response was defined as the number of days from the day a participants received the first dose of guadecitabine (cycle 1 day 1 {C1D1}) to the first day of response. Composite complete response rate (CRc = CR + CRp + CRi), which is an overall complete response assessment including CR, CR with incomplete platelet recovery (CRp) and CR with incomplete blood count recovery (CRi). CRc rate, was defined as the number of participants who achieved a response status of CR, CRp, or CRi divided by the total number of participants included in the efficacy dataset. The CR rate is defined as the number of participants whose best response is CR divided by the total number of participants included in the efficacy dataset.
Time Frame: At end of each Cycle of 28 days (Up to approximately 38 months)
Population: Efficacy analysis set included regimen 1, 2A and 2B, r/r AML and TN AML participants who received at least one dose of study drug. Data is reported for responders in this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 3 | 2 | 0
days | 106.0 [106 to 147] | 55.5 [27 to 84] |

14. Secondary Outcome: Dose Expansion Phase- r/r MDS, TN MDS: Time to Response
Description: Time to response was defined as the number of days from the day a participants received the first dose of guadecitabine (C1D1) to the first day of response. CR:normal peripheral counts with persistent granulocyte count ≥1.0×10^9/L, platelet count ≥100×10^9/L and normal bone marrow (BM) with persistent marrow blasts ≤5%; persistent dysplasia was noted. PR:normal peripheral counts with granulocyte count ≥1.0×10^9/L and platelet count ≥100 ×10^9/L and normal BM with marrow blasts >5% but were reduced by 50% or more. mCR:reduction of BM blasts to ≤5% without normalization of peripheral counts. HI is divided as erythroid response(HI-E): hemoglobin increase ≥1.5 g/dL or RBC transfusion independence, platelet response (HI-P): absolute increase of platelet count from <20 to >20×10^9/L by at least 100%,/if more than 20×10^9/L, by absolute increase of 30×10^9/L, neutrophil response (HI-N): granulocyte increase ≥100%, by an absolute increase ≥0.5×10^9/L.
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included r/r MDS and TN MDS participants who received at least one dose of study drug. Overall number of participants analysed are the participants with response. Number analyzed is number of participants with response.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 6 | 12 | 12 | 11
days
  CR+PR+mCR: number analyzed (Participants) | 5 | 12 | 7 | 11
  CR+PR+mCR | 27.0 [25 to 512] | 68.0 [23 to 189] | 196.0 [24 to 245] | 133 [47 to 392]
  HI: number analyzed (Participants) | 6 | 9 | 12 | 9
  HI | 108.0 [5 to 173] | 58.0 [27 to 277] | 64.5 [0 to 364] | 49.0 [27 to 119]

15. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) Assessed Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: DLT was defined using CTCAE v4.0. Toxicities were considered related to SGI-110 if it cannot be explained by underlying disease, intercurrent illness or concomitant medications. Any related Grade 3 or 4 non-hematologic toxicity except Grade 3 or 4 nausea/vomiting that is controllable by anti-emetics or diarrhea controllable by optimal therapy. Grade 3 laboratory investigations other than serum creatinine, bilirubin, AST or ALT were not considered a DLT unless they are associated with clinical manifestations. Study-drug related Grade 4 thrombocytopenia and Febrile neutropenia that was not present at study entry, and not resolve within 7 days, and is not related to underlying disease. Prolonged myelosuppression or pancytopenia with hypocellular bone marrow and no marrow blasts lasting for 6 weeks or more that is not related to disease progression. Any toxicity that results in treatment delays of > 4 weeks. Data is reported for any AE occurring during Cycle 1 (each cycle = 28 days).
Time Frame: Cycle 1 (each cycle = 28 days)
Population: Safety analysis set included data from regimen 1, 2A and 2B participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 44 | 34 | 15
Participants | 2 | 0 | 0

16. Secondary Outcome: Dose Escalation and Dose Expansion Phases- r/r AML, TN AML, r/r MDS, TN MDS: Number of Participants With At Least One Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent AEs are defined as events that first occurred or worsened after the first dose of study drug given on C1D1 until 30 days after the last dose of study treatment or the start of an alternative anti-cancer treatment for MDS/CMML and subsequent AML, whichever occurs first, with the following exceptions: events that occurred after 30 days beyond the last dose of study treatment or the start of an alternative anti-cancer treatment for MDS/CMML and subsequent AML was considered treatment-emergent if the events are both serious and related to the study treatment.
Time Frame: From first dose of study drug up 30 days post treatment (up to approximately 46 months)
Population: Safety data set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 44 | 34 | 15 | 24 | 26 | 53 | 24 | 27 | 52 | 26 | 27 | 27 | 22
Participants | 44 | 34 | 15 | 24 | 26 | 53 | 24 | 27 | 52 | 26 | 27 | 27 | 22

17. Secondary Outcome: Dose Escalation and DE Phases- r/r AML, TN AML, r/r MDS, TN MDS: Number of Participants With Abnormal Laboratory Values Reported as Adverse Events
Time Frame: From first dose of study drug up 30 days post treatment (up to approximately 46 months)
Population: Safety data set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly: Participants received starting dose of guadecitabine 6 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle. The dose was subsequently increased to 18, 36, 60, 90, 125 mg/m^2 for subsequent cycles until development of toxicity or disease progression.
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 44 | 34 | 15 | 24 | 26 | 53 | 24 | 27 | 52 | 26 | 27 | 27 | 22
Participants
  Alanine Aminotransferase Increased | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 6 | 0 | 2 | 1 | 0
  Hypoalbuminaemia | 6 | 3 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 2 | 2 | 1
  Blood Alkaline Phosphatase Increased | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Blood Alkaline Phosphatase Decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase Increased | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 1
  Blood Creatinine Increased | 3 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 4 | 0 | 2 | 2 | 1
  Blood Creatinine Decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Magnesium Increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Potassium Increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 0
  Hyperbilirubinaemia | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0

18. Secondary Outcome: Dose Escalation: Maximum Observed Plasma Concentration (Cmax ) of SGI-110 and Decitabine
Time Frame: Days 1, 5 and 8
Population: Pharmacokinetic (PK) analysis set included all available plasma concentrations and PK parameters for guadecitabine and decitabine for participants who received study drug. Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dose Escalation: Regimen 1: Once Daily - 3 mg/m^2: Participants received starting dose of guadecitabine 3 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 1: Once Daily - 9 mg/m^2: Participants received starting dose of guadecitabine 9 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 1: Once Daily - 18 mg/m^2: Participants received starting dose of guadecitabine 18 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 1: Once Daily - 36 mg/m^2: Participants received starting dose of guadecitabine 36 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 1: Once Daily - SGI-110 - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 1: Once Daily - 90 mg/m^2: Participants received starting dose of guadecitabine 90 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 1: Once Daily - 125 mg/m^2: Participants received starting dose of guadecitabine 125 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Weekly- 6 mg/m^2: Participants received starting dose of guadecitabine 6 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Weekly- 18 mg/m^2: Participants received starting dose of guadecitabine 18 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: 10. Regimen 2A: Once Weekly- 36 mg/m^2: Participants received starting dose of guadecitabine 36 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Weekly - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Weekly - 90 mg/m^2: Participants received starting dose of guadecitabine 90 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Weekly - 125 mg/m^2: Participants received starting dose of guadecitabine 125 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2B: Twice Weekly - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, twice weekly on Days 1, 4, 8, 11, 15 and 18 of a 28-day cycle.
Arm/Group | Dose Escalation: Regimen 1: Once Daily - 3 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 9 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 18 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 36 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - SGI-110 - 60 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 90 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 125 mg/m^2 | Dose Escalation: Regimen 2A: Once Weekly- 6 mg/m^2 | Dose Escalation: Regimen 2A: Once Weekly- 18 mg/m^2 | Dose Escalation: 10. Regimen 2A: Once Weekly- 36 mg/m^2 | Dose Escalation: Regimen 2A: Once Weekly - 60 mg/m^2 | Dose Escalation: Regimen 2A: Once Weekly - 90 mg/m^2 | Dose Escalation: Regimen 2A: Once Weekly - 125 mg/m^2 | Dose Escalation: Regimen 2B: Twice Weekly - 60 mg/m^2
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 7 | 6 | 12 | 6 | 3 | 6 | 4 | 7 | 6 | 7
ng/mL
  SGI-110: Day 1: number analyzed (Participants) | 4 | 4 | 5 | 6 | 7 | 6 | 12 | 6 | 3 | 6 | 4 | 6 | 6 | 7
  SGI-110: Day 1 | 6.69 (72.9) | 19.1 (43.5) | 45.7 (57.9) | 106 (129) | 121 (31.9) | 155 (34.6) | 178 (46.2) | 11.7 (65.7) | 37.4 (73.4) | 61.9 (44.5) | 101 (51.0) | 100 (30.2) | 219 (36.5) | 106 (29.9)
  SGI-110: Day 5: number analyzed (Participants) | 4 | 4 | 5 | 6 | 5 | 6 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SGI-110: Day 5 | 11.1 (65.8) | 30.7 (42.5) | 45.2 (43.4) | 72.7 (41.1) | 120 (31.7) | 205 (34.9) | 173 (36.7) |  |  |  |  |  |  |
  SGI-110: Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 6 | 4 | 7 | 6 | 0
  SGI-110: Day 8 |  |  |  |  |  |  |  | 10.7 (60.7) | 18.1 (99.3) | 66.3 (63.8) | 107 (40.0) | 118 (27.8) | 187 (40.9) |
  Decitabine: Day 1: number analyzed (Participants) | 4 | 4 | 5 | 6 | 7 | 6 | 12 | 6 | 3 | 6 | 4 | 6 | 6 | 7
  Decitabine: Day 1 | 1.27 (30.5) | 2.54 (18.5) | 8.18 (56.9) | 13.9 (60.4) | 23.7 (79.8) | 42.0 (40.0) | 61.5 (37.4) | 3.05 (48.4) | 8.20 (52.7) | 17.1 (55.9) | 16.7 (47.0) | 30.1 (41.3) | 65.9 (50.0) | 26.1 (83.2)
  Decitabine: Day 5: number analyzed (Participants) | 4 | 4 | 5 | 6 | 5 | 6 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Decitabine: Day 5 | 1.67 (54.7) | 3.52 (27.4) | 10.3 (65.1) | 16.7 (37.6) | 22.7 (69.9) | 53.6 (37.4) | 59.1 (30.5) |  |  |  |  |  |  |
  Decitabine: Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 6 | 4 | 7 | 6 | 0
  Decitabine: Day 8 |  |  |  |  |  |  |  | 2.78 (43.8) | 6.92 (79.5) | 12.7 (41.8) | 19.0 (55.8) | 35.0 (45.4) | 53.2 (39.5) |

19. Secondary Outcome: Dose Escalation: Minimum Observed Plasma Concentration (Cmin)
Time Frame: Days 5 and 8
Population: PK analysis set included all available plasma concentrations and PK parameters for guadecitabine and decitabine for participants who received study drug. Overall number of participants analyzed are the number of participants available for analysis. Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dose Escalation: Regimen 1: Once Daily - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, daily from Days 1-5 of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Daily - 6 mg/m^2: Participants received starting dose of guadecitabine 6 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Daily - 18 mg/m^2: Participants received starting dose of guadecitabine 18 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Daily - 36 mg/m^2: Participants received starting dose of guadecitabine 36 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Daily - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Daily - 90 mg/m^2: Participants received starting dose of guadecitabine 90 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2A: Once Daily - 125 mg/m^2: Participants received starting dose of guadecitabine 125 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2B: Once Daily - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, twice weekly on Days 1, 4, 8, 11, 15 and 18of a 28-day cycle.
Arm/Group | Dose Escalation: Regimen 1: Once Daily - 3 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 9 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 18 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 36 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 60 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 90 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 125 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 6 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 18 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 36 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 60 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 90 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 125 mg/m^2 | Dose Escalation: Regimen 2B: Once Daily - 60 mg/m^2
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 7 | 6 | 12 | 5 | 3 | 6 | 4 | 8 | 6 | 0
ng/mL
  SGI-110: Day 5: number analyzed (Participants) | 4 | 4 | 5 | 6 | 7 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SGI-110: Day 5 | NA (NA) — Data could not be estimable as the values were below lower limit of quantitation (LLOQ) | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. |  |  |  |  |  |  |
  SGI-110: Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 6 | 4 | 8 | 6 | 0
  SGI-110: Day 8 |  |  |  |  |  |  |  | NA (224) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (200) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. | NA (NA) — Data could not be estimable as the values were below LLOQ. |

20. Secondary Outcome: Dose Escalation: Area Under the Curve to Infinity (AUC0-inf)
Time Frame: Days 1, 5 and 8
Population: Pharmacokinetic (PK) analysis set included all available plasma concentrations and PK parameters for guadecitabine and decitabine for participants who received study drug. Overall number of participants analyzed are the number of participants available for analysis. Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Dose Escalation: 10. Regimen 2A: Once Daily - 36 mg/m^2: Participants received starting dose of guadecitabine 36 mg/m^2, SC, once weekly on Days 1, 8 and 15, SC of a 28-day cycle.
- Dose Escalation: Regimen 2B: Once Daily - 60 mg/m^2: Participants received starting dose of guadecitabine 60 mg/m^2, SC, twice weekly on Days 1, 4, 8, 11, 15 and 18 of a 28-day cycle.
Arm/Group | Dose Escalation: Regimen 1: Once Daily - 3 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 9 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 18 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 36 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - SGI-110 - 60 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 90 mg/m^2 | Dose Escalation: Regimen 1: Once Daily - 125 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 6 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 18 mg/m^2 | Dose Escalation: 10. Regimen 2A: Once Daily - 36 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 60 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 90 mg/m^2 | Dose Escalation: Regimen 2A: Once Daily - 125 mg/m^2 | Dose Escalation: Regimen 2B: Once Daily - 60 mg/m^2
Number analyzed (Participants) | 3 | 4 | 5 | 6 | 7 | 6 | 12 | 6 | 2 | 6 | 5 | 6 | 7 | 6
ng*hr/mL
  SGI-110: Day 1: number analyzed (Participants) | 3 | 4 | 5 | 5 | 7 | 6 | 12 | 6 | 2 | 6 | 5 | 6 | 6 | 6
  SGI-110: Day 1 | 12.1 (71.5) | 45.2 (23.9) | 102 (42.7) | 211 (55.8) | 410 (25.8) | 528 (26.8) | 648 (31.3) | 21.4 (65.4) | 99.8 (25.2) | 182 (19.5) | 327 (48.9) | 331 (23.1) | 636 (40.2) | 328 (38.4)
  SGI-110: Day 5: number analyzed (Participants) | 2 | 4 | 5 | 6 | 5 | 6 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SGI-110: Day 5 | 26.5 (5.87) | 63.5 (13.7) | 112 (29.8) | 226 (35.0) | 354 (13.8) | 423 (46.0) | 658 (26.9) |  |  |  |  |  |  |
  SGI-110: Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 5 | 4 | 6 | 7 | 0
  SGI-110: Day 8 |  |  |  |  |  |  |  | 17.9 (42.1) | 58.0 (15.0) | 227 (50.5) | 371 (15.2) | 383 (27.4) | 675 (45.1) |

21. Secondary Outcome: Dose Escalation and DE Phase- r/r MDS, TN MDS: Time to AML or Death
Description: Time to AML or death was defined as the number of days from the date the subject received the first dose of guadecitabine (C1D1) to the date of death or the date of MDS/ chronic myelomonocytic leukemia (CMML) progression to AML, whichever occurred earlier. Time to AML or death was evaluated using the Kaplan-Meier method, with the time censored on the last date of contact if a participant was still alive without progression to AML.
Time Frame: At end of each Cycle of 28 days (Up to approximately 38 months)
Population: Efficacy analysis set included Regimen 1, 2A, 2B, r/r MDS and TN MDS participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 44 | 35 | 15 | 26 | 27 | 27 | 22
days | 244.5 [165.0 to 581.0] | 275.0 [197.0 to 585.0] | 373.0 [212.0 to NA] — Upper limit of full range was not estimable due to insufficient number of participants with events. | 273 [164.0 to 622.0] | 276 [175.0 to 436.0] | 680 [402.0 to 848.0] | 542.5 [224.0 to NA] — Upper limit of full range was not estimable due to insufficient number of participants with events.

22. Secondary Outcome: Dose Escalation and DE Phases- r/r AML, TN AML, r/r MDS, TN MDS: Overall Survival
Description: OS was defined as the number of days from the day the participant received the first dose of guadecitabine to the date of death (regardless of cause).
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 44 | 35 | 15 | 50 | 53 | 0 | 0 | 0 | 0 | 26 | 27 | 27 | 22
days | 124 [82.0 to 181.0] | 186.5 [115.0 to 236.0] | 212.0 [111.0 to 304.0] | 172 [142.0 to 254.0] | 214 [169.0 to 269.0] |  |  |  |  | 273 [199.0 to 622.0] | 370 [253.0 to 447.0] | 771 [460.0 to 1017.0] | 558 [269.0 to NA] — Upper limit of full range was not estimable due to insufficient number of participants with events.

23. Secondary Outcome: Dose Escalation: Number of Participants Achieving Blood and Platelet Transfusions
Time Frame: Cycle 1, Day 1 through 30 days after the last dose of study drug (up to approximately 46 months)
Population: Efficacy analysis set included all participants who received at least one dose of study drug. Overall number of participants are the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly
Number analyzed (Participants) | 23 | 16 | 8
percentage of participants
  (Maintaining/achieving platelet transfusion independence): number analyzed (Participants) | 19 | 16 | 6
  (Maintaining/achieving platelet transfusion independence) | 100 | 89 | 75
  (Maintaining/achieving RBC transfusion independence): number analyzed (Participants) | 23 | 15 | 8
  (Maintaining/achieving RBC transfusion independence) | 100 | 79 | 89

24. Secondary Outcome: DE Phase- r/r AML, TN AML: Percentage of Participants With Cr, CRp and PR
Description: CR is defined absolute neutrophil count (ANC) >1.0×109/L, Platelets ≥100×109/L, independence from RBC and platelet transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRp is defined ANC >1.0×10^9/L, Platelets <100×10^9/L, independence from RBC transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRi is defined as ANC <1.0×10^9/L, no myeloblasts and <5% myeloblasts in bone marrow. PR is defined as ANC >1.0×10^9/L, Platelets ≥100×10^9/L, no myeloblasts and Decrease of ≥50% in myeloblasts to level of 5% to 25% in bone marrow.
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included r/r AML and TN AML participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day)
Number analyzed (Participants) | 24 | 26 | 53 | 24 | 27 | 52
percentage of participants
  CR | 8.3 | 7.7 | 18.9 | 37.5 | 40.7 | 32.7
  CRi | 4.2 | 11.5 | 3.8 | 16.7 | 11.1 | 7.7
  CRp | 0 | 0 | 7.5 | 0 | 7.4 | 9.6
  PR | 0 | 0 | 0 | 4.2 | 3.7 | 1.9

25. Secondary Outcome: DE Phase- r/r MDS, TN MDS: Percentage of Participants With CR, PR, mCR and HI
Description: CR is defined ANC >1.0×109/L, Platelets ≥100×109/L, independence from RBC and platelet transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRp is defined ANC >1.0×10^9/L, Platelets <100×10^9/L, independence from RBC transfusions over the past week, no myeloblasts and <5% myeloblasts in bone marrow. CRi is defined as ANC <1.0×10^9/L, no myeloblasts and <5% myeloblasts in bone marrow. PR is defined as ANC >1.0×10^9/L, Platelets ≥100×10^9/L, no myeloblasts and Decrease of ≥50% in myeloblasts to level of 5% to 25% in bone marrow.
Time Frame: At end of each Cycle of 28 days (Up to approximately 45 months)
Population: Efficacy analysis set included r/r MDS and TN MDS participants who received at least one dose of study drug. Overall number of participants are the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 26 | 27 | 27 | 22
percentage of participants
  CR+PR+mCR | 19 | 44 | 26 | 50
  HI | 23 | 33 | 44 | 41

26. Secondary Outcome: DE Phase- r/r MDS, TN MDS: Number of Participants Achieving Blood Transfusion Independence for 8 or 16-weeks
Description: Transfusion dependence at baseline was defined as any transfusion within 4 weeks of the first study dose (C1D1) with C1D1 transfusion counted, assuming it was always done before dosing. Transfusion independence after treatment was defined as no transfusion within an 8-week or 16-week period between C1D1 and last treatment date + 30 days.
Time Frame: Weeks 8 and 16
Population: Efficacy analysis set included r/r MDS and TN MDS participants who received at least one dose of study drug. Overall Number of Participants Analyzed are those who were dependent on RBC transfusions at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 16 | 18 | 15 | 9
Participants
  RBC Independence for Week 8 | 1 | 4 | 6 | 4
  RBC Independence for Week 16 | 0 | 3 | 5 | 1

27. Secondary Outcome: DE Phase- r/r MDS, TN MDS: Number of Participants Achieving Platelet Transfusion Independence for 8 or 16-weeks
Description: as for outcome 26
Time Frame: Weeks 8 and 16
Population: Efficacy analysis set included r/r MDS and TN MDS participants who received at least one dose of study drug. Overall Number of Participants Analyzed are those who were dependent on platelet transfusions at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
Number analyzed (Participants) | 6 | 10 | 7 | 5
Participants
  Platelet Independence for Week 8 | 0 | 5 | 3 | 3
  Platelet Independence for Week 16 | 0 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days post study treatment (up to 46 months)
Description: All-cause mortality is reported for all enrolled participants. Serious adverse events are reported for safety set which included data from all participants who received at least one dose of study drug. Reconciling the >=5% adverse event data collected in multiple cohorts in trials conducted approximately 10 years ago cannot be provided as a single comprehensive data set, therefore no data is available to report for this safety section.
Arm/Group | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day)
All-Cause Mortality (participants affected / at risk) | 5/44 | 4/35 | 0/15 | 4/25 | 3/28 | 10/55 | 4/24 | 7/27 | 11/52 | 2/26 | 4/27 | 1/27 | 2/22
Serious Adverse Events (participants affected / at risk) | 33/44 | 28/34 | 8/15 | 19/24 | 21/26 | 44/53 | 21/24 | 24/27 | 45/52 | 17/26 | 22/27 | 17/27 | 17/22
Other Adverse Events (participants affected / at risk) | 44/44 | 34/34 | 15/15 | 24/24 | 26/26 | 53/53 | 24/24 | 27/27 | 52/52 | 26/26 | 27/27 | 27/27 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily (N=44) | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly (N=34) | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly (N=15) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) (N=24) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) (N=26) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) (N=53) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) (N=24) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) (N=27) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) (N=52) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) (N=26) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) (N=27) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) (N=27) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day) (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 11 | 5 | 9 | 10 | 28 | 12 | 15 | 25 | 9 | 11 | 7 | 9
Pneumonia (Infections and infestations) | 15 | 8 | 3 | 5 | 9 | 17 | 4 | 10 | 16 | 4 | 10 | 7 | 4
Sepsis (Infections and infestations) | 8 | 6 | 2 | 2 | 2 | 11 | 2 | 6 | 14 | 2 | 4 | 0 | 3
Cellulitis (Infections and infestations) | 3 | 3 | 0 | 4 | 0 | 5 | 2 | 2 | 1 | 0 | 2 | 2 | 4
Bacteraemia (Infections and infestations) | 3 | 2 | 0 | 3 | 3 | 3 | 2 | 3 | 3 | 1 | 4 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 2
Anorectal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Regimen 1 - Guadecitabine 3 mg/m^2 Daily (N=44) | Dose Escalation: Regimen 2A - Guadecitabine 6 mg/m^2 Once Weekly (N=34) | Dose Escalation: Regimen 2B - Guadecitabine 60 mg/m^2 Twice Weekly (N=15) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (5-Day) (N=24) | Dose Expansion: r/r AML Guadecitabine 90 mg/m^2 (5-Day) (N=26) | Dose Expansion: r/r AML Guadecitabine 60 mg/m^2 (10-Day) (N=53) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (5-Day) (N=24) | Dose Expansion: TN AML Guadecitabine 90 mg/m^2 (5-Day) (N=27) | Dose Expansion: TN AML Guadecitabine 60 mg/m^2 (10-Day) (N=52) | Dose Expansion: r/r MDS Guadecitabine 60 mg/m^2 (5-Day) (N=26) | Dose Expansion: r/r MDS Guadecitabine 90 mg/m^2 (5-Day) (N=27) | Dose Expansion: TN MDS Guadecitabine 60 mg/m^2 (5-Day) (N=27) | Dose Expansion: TN MDS Guadecitabine 90 mg/m^2 (5-Day) (N=22)
Anaemia (Blood and lymphatic system disorders) | 11 | 8 | 5 | 6 | 6 | 28 | 11 | 10 | 14 | 15 | 13 | 11 | 13
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 8 | 0 | 1 | 4 | 0 | 2 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 5 | 3 | 0 | 0 | 0 | 5 | 7 | 16 | 1 | 0 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 4 | 6 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 4 | 1 | 3 | 4 | 4 | 6 | 6 | 2 | 2 | 4 | 5 | 4
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 2 | 4 | 3 | 3 | 15 | 9 | 12 | 18 | 14 | 12 | 11 | 14
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 6 | 4 | 6 | 5 | 26 | 13 | 12 | 24 | 14 | 14 | 9 | 12
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 1 | 0 | 1 | 4 | 1 | 2 | 3 | 2 | 1 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 3 | 5 | 0 | 1 | 2 | 2 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 4 | 3 | 0 | 2 | 0 | 5 | 0 | 1 | 6 | 3 | 1 | 0 | 1
Auricular swelling (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 3 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 2 | 4 | 1 | 3 | 5 | 1 | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 0 | 4 | 2 | 12 | 4 | 7 | 5 | 3 | 0 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 3 | 2 | 2 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 6 | 2 | 5 | 9 | 22 | 12 | 14 | 32 | 5 | 6 | 10 | 12
Diarrhoea (Gastrointestinal disorders) | 22 | 11 | 2 | 6 | 9 | 28 | 10 | 12 | 31 | 7 | 15 | 10 | 7
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 2 | 1 | 0 | 3 | 7 | 4 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 4 | 6 | 1 | 3 | 5 | 3 | 7 | 2 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 2 | 3 | 3 | 2 | 2 | 1 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 3 | 1 | 2 | 0
Gingival erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 1 | 5 | 0 | 4 | 4 | 2 | 3 | 1 | 1
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 1 | 2 | 0 | 4 | 3 | 2 | 3 | 3 | 1
Nausea (Gastrointestinal disorders) | 12 | 9 | 0 | 6 | 5 | 31 | 11 | 13 | 26 | 10 | 8 | 8 | 12
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 3 | 2 | 0 | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 6 | 3 | 3 | 1 | 4 | 19 | 4 | 9 | 15 | 2 | 11 | 3 | 7
Stomatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 5 | 0 | 5 | 1 | 21 | 6 | 5 | 16 | 3 | 3 | 7 | 9
Asthenia (General disorders) | 4 | 7 | 3 | 3 | 3 | 8 | 5 | 7 | 19 | 5 | 2 | 5 | 6
Catheter site erythema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 3 | 1 | 0 | 0 | 0 | 4 | 2 | 1 | 4 | 0 | 1 | 0 | 0
Chills (General disorders) | 3 | 5 | 2 | 0 | 2 | 5 | 2 | 3 | 6 | 0 | 2 | 1 | 6
Device occlusion (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 11 | 9 | 7 | 7 | 9 | 26 | 11 | 10 | 21 | 11 | 10 | 12 | 9
Gait disturbance (General disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Infusion site induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Injection site haematoma (General disorders) | 1 | 2 | 0 | 3 | 2 | 5 | 2 | 6 | 1 | 1 | 6 | 5 | 5
Injection site haemorrhage (General disorders) | 1 | 1 | 2 | 2 | 2 | 2 | 3 | 5 | 0 | 0 | 0 | 1 | 2
Injection site mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 1 | 0 | 1 | 2 | 5 | 2 | 5 | 6 | 1 | 4 | 8 | 4
Injection site pain (General disorders) | 11 | 11 | 9 | 7 | 9 | 18 | 11 | 16 | 6 | 8 | 9 | 11 | 12
Injection site reaction (General disorders) | 2 | 1 | 2 | 1 | 0 | 6 | 2 | 2 | 7 | 3 | 1 | 4 | 4
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 3 | 2 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 12 | 0 | 1 | 1 | 2
Oedema peripheral (General disorders) | 11 | 9 | 3 | 3 | 4 | 16 | 8 | 10 | 15 | 8 | 5 | 4 | 4
Pain (General disorders) | 0 | 1 | 0 | 0 | 2 | 5 | 5 | 2 | 13 | 1 | 2 | 1 | 2
Pyrexia (General disorders) | 7 | 8 | 1 | 3 | 4 | 8 | 5 | 6 | 9 | 1 | 7 | 1 | 3
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune system disorder (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute haemorrhagic conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 5 | 2 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 4 | 0 | 2 | 4 | 0 | 2 | 1 | 1
Cellulitis (Infections and infestations) | 7 | 4 | 0 | 3 | 3 | 8 | 3 | 3 | 14 | 1 | 2 | 4 | 5
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 2 | 2 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 0 | 0 | 2 | 6 | 1 | 0 | 3 | 1 | 2 | 0 | 1
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 4 | 1 | 2 | 2 | 15 | 3 | 5 | 8 | 3 | 5 | 2 | 2
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Streptococcal urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 1 | 1 | 1 | 3 | 1 | 4 | 4 | 1 | 5 | 4 | 4
Urethritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 5 | 1 | 0 | 0 | 8 | 3 | 2 | 6 | 1 | 3 | 3 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 4 | 3 | 0 | 1 | 8 | 8 | 5 | 11 | 9 | 5 | 7 | 6
Excoriation (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 5 | 2 | 2 | 10 | 4 | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Underdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 6 | 0 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0 | 0 | 1 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 0 | 0 | 2 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 4 | 0 | 2 | 2 | 1
Blood fibrinogen increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram qt prolonged (Investigations) | 1 | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Fibrinolysis increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0
Occult blood positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 2 | 3 | 1 | 0 | 1 | 7 | 5 | 1 | 3 | 3 | 2 | 3 | 2
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 4 | 4 | 4 | 6 | 25 | 8 | 14 | 20 | 8 | 8 | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 2 | 2 | 1 | 5
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 5 | 0 | 2 | 1 | 1 | 1 | 5 | 3 | 0 | 2 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 2 | 0 | 1 | 1 | 1 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 | 6 | 4 | 2 | 1 | 3 | 1 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 3 | 2 | 2 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 3 | 0 | 0 | 1 | 7 | 1 | 1 | 3 | 0 | 2 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 0 | 2 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 9 | 1 | 9 | 11 | 25 | 9 | 14 | 27 | 2 | 8 | 6 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 6 | 2 | 4 | 8 | 27 | 6 | 8 | 23 | 4 | 4 | 9 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 6 | 1 | 0 | 2 | 5 | 3 | 3 | 8 | 1 | 3 | 6 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4 | 0 | 4 | 4 | 5 | 2 | 6 | 6 | 1 | 2 | 2 | 1
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 0 | 1 | 0 | 6 | 3 | 4 | 8 | 5 | 2 | 4 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 2 | 1 | 10 | 6 | 3 | 12 | 2 | 3 | 6 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0 | 0 | 5 | 0 | 1 | 2 | 0 | 1 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 5 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 3 | 2 | 5 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 4 | 3 | 0 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 1 | 0 | 4 | 2 | 2 | 3 | 2 | 0 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 1 | 0 | 6 | 3 | 0 | 4 | 7 | 3 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2 | 2 | 2 | 5 | 2 | 3 | 7 | 2 | 3 | 8 | 5
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Consciousness fluctuating (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 3 | 2 | 0 | 0 | 0 | 6 | 8 | 14 | 7 | 5 | 5 | 4
Dysgeusia (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 3 | 1 | 4 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 6 | 3 | 5 | 3 | 13 | 6 | 6 | 8 | 4 | 6 | 3 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pachymeningitis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 1 | 2 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 0 | 0 | 1 | 0
Viith nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 3 | 1 | 0 | 2 | 8 | 2 | 1 | 14 | 3 | 1 | 1 | 2
Depression (Psychiatric disorders) | 5 | 1 | 1 | 0 | 0 | 11 | 5 | 3 | 5 | 3 | 1 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 8 | 0 | 4 | 2 | 10 | 6 | 5 | 6 | 6 | 6 | 5 | 8
Mental status changes (Psychiatric disorders) | 3 | 1 | 0 | 3 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 6 | 0 | 0 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 4 | 1 | 2 | 0
Renal failure (Renal and urinary disorders) | 5 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 3 | 1 | 1 | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 1 | 0 | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 2 | 4 | 7 | 22 | 9 | 6 | 20 | 8 | 10 | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 3 | 6 | 4 | 9 | 6 | 12 | 26 | 4 | 6 | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 3 | 4 | 6 | 8 | 3 | 7 | 13 | 6 | 7 | 5 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 5 | 1 | 0 | 3 | 0 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 0 | 0 | 1 | 8 | 0 | 0 | 3 | 3 | 6 | 3 | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 3 | 3 | 9 | 2 | 5 | 13 | 2 | 3 | 4 | 4
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2 | 3 | 1 | 2 | 1 | 8 | 1 | 2 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 4 | 1 | 2 | 7 | 4 | 3 | 2 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 0 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 4 | 0 | 3 | 1 | 2 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 2 | 2 | 0 | 2 | 5 | 0 | 0 | 4 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 0 | 4 | 0 | 3 | 11 | 1 | 1 | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 4 | 6 | 1 | 0 | 0 | 3 | 3 | 2 | 9 | 3 | 3 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 2 | 4 | 0 | 1 | 8 | 2 | 3 | 2 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 1 | 3 | 3 | 1 | 6 | 2 | 5 | 5 | 6 | 4 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 1 | 1 | 3 | 3 | 0 | 6 | 1 | 2 | 2 | 4
Pruritus generalised (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 9 | 3 | 1 | 2 | 11 | 1 | 4 | 11 | 2 | 4 | 9 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 1 | 3 | 3 | 1 | 5 | 1 | 1 | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vagotomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 5 | 2 | 2 | 1 | 2 | 1
Hypertension (Vascular disorders) | 1 | 3 | 2 | 0 | 2 | 5 | 1 | 2 | 0 | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 10 | 4 | 2 | 4 | 5 | 10 | 3 | 3 | 10 | 3 | 4 | 2 | 2
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 11 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
External ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Scleral disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scotoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 2 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bk virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-barr viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fusarium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterium kansasii infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sweating fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheostomy infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 3
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 5 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum culture (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin i increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 3 | 3 | 1 | 10 | 1 | 0 | 0 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epstein-barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 2 | 4 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vulvar erosion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Enterostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Maxillofacial operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 5 | 0 | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conjunctival pallor (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Eyelid disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pupillary disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scleral pigmentation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site joint redness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Genital abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspergillus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Enterobacter test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alkalosis hypochloraemic (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 10 | 0 | 0 | 0 | 0
Delirium febrile (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 2 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoperfusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival discolouration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crepitations (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site joint swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis c (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suture related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Floating patella (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anhedonia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cutis laxa (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palpable purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No